CLINICAL TRIAL: NCT01008501
Title: Genetic Studies in Gestational Trophoblastic Disease
Brief Title: Study of the Genetic and Epigenetic Causes of Recurrent Hydatidiform Moles
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ignatia Van den Veyver, Professor, Baylor College of Medicine
Other Study IDs: BCM Hydatidiform Mole H7345
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hydatidiform Moles
Keywords: hydatidiform moles; complete hydatidiform moles; partial hydatidiform moles; Molar pregnancy; NLRP7; pregnancy wastage; imprinting; sporadic hydatidiform moles; recurrent hydatidiform moles
MeSH Terms: conditions — Hydatidiform Mole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lymphoblast DNA; tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental: Individuals with recurrent or sporadic hydatidiform moles and their first-degree family members. Sometimes additional family members are also enrolled.

SUMMARY:
The researchers' laboratory is studying a rare class of highly recurrent hydatidiform moles. These are usually complete hydatidiform moles (CHM), but sometimes they are partial hydatidiform moles PHM). With sporadic moles, the difference between CHMs and PHMs is that with CHMS, there is not typically an embryo or fetus at the time of diagnosis but with a PHM there may be a fetus. Also, CHMs have 46 chromosomes in each cell. While this is the number of chromosomes that should be found, the problem is that all the chromosomes come from the father. Normally, half the chromosomes should come from the mother and half should come from the father. Unlike CHMs, PHMs have 69 chromosomes. This means that PHMs have three copies of each chromosome when they should only have two. The extra copy comes from the father.

The researchers' study focuses on moles that are genetically different from these sporadic moles in that they have 23 chromosomes from the mother and 23 chromosomes from the father - just like a normally developing pregnancy. These are called biparental moles because the mutation that causes the mole comes from both parents. This mutation occurs in a gene called NLRP7. The researchers' team is working to understand how mutations in NLRP7 leads to CHMs and how these mutations may lead to other types of pregnancy loss. The researchers are also trying to discover other genetic and epigenetic factors that may lead to moles.

DETAILED DESCRIPTION:
Hydatidiform mole (HM) is the product of an aberrant human pregnancy in which there is abnormal embryonic development and abnormal proliferation of placental villi. The incidence of HM varies between ethnic groups, and occurs in 1 in every 1500 pregnancies in the USA. All HM cases are sporadic except for extremely rare familial cases. The exact mechanisms leading to molar pregnancies are not known. Hydatidiform moles are classified based on histology and karyotype data into two types:

complete hydatidiform moles (CHM) and partial hydatidiform moles (PHM). The complete forms are characterized by general trophoblastic proliferation and absence of an embryo and amniotic membranes. In most of the cases, CHM have a diploid genome, and are androgenetic with two identical sets of paternal chromosomes. Partial hydatidiform moles are characterized by focal trophoblastic proliferation. Embryos and amniotic membranes are usually present in these molar pregnancies. Partial hydatidiform moles are mostly triploid with two sets of paternal chromosomes and one set of maternal chromosomes. The comparison of findings in androgenetic CHM and PHM indicate that both maternally (under) expressed and paternally (over) expressed genes play a role in the pathophysiology of molar pregnancies. Very few genetic studies have been performed on molar pregnancies or the patients who carry these pregnancies. A few studies have looked at the over- or underexpression of genes that may play a role in the progression or invasiveness of hydatidiform moles; however none have addressed the underlying genetic etiology. We have been able to study an inbred family of which several female members have had recurrent hydatidiform moles and have now genetically mapped the defective gene responsible for the molar pregnancies in this family. We then worked towards refined characterization of the genetic locus containing the mutated gene and analysis of candidate genes in this region for mutations leading to molar pregnancy. Because the hydatidiform moles in these patients have abnormal genetic imprinting, we believe that this candidate gene is important for establishment of genetic imprinting in the maternal germline. Recently, another group of investigators studying this condition identified mutations in a gene, NALP7 (now renamed to NLRP7), in some of the affected women. We confirmed this in other subjects studied by us. This is the first identified gene, but there is genetic heterogeneity and other genes still remain to be found. In addition, the normal function of this gene in reproduction and how it leads to recurrent moles when mutated remains to be determined. To study both of these, it will be very important to collect as many molar pregnancy tissue samples as possible, as well as blood samples and/or other non-invasively obtained samples, such as buccal swabs and saliva, from affected patients and their families. Recent evidence suggests that mutations in NLRP7 might cause other forms of reproductive failure, such as triploid spontaneous abortions. It has further been proposed that the mutation status of NLRP7 in women with recurrent reproductive loss is an important predictor of the outcome of Assisted Reproductive Technologies. Therefore, we are carrying out mutation analysis of NLRP2 and NLRP7 in women with unexplained infertility and other forms of reproductive failure.

ELIGIBILITY:
Inclusion Criteria:

* Personal or family history of recurrent moles or a sporadic mole
* Presence of a mutation in NLRP7

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have had sporadic or recurrent hydatidiform moles and their first degree relatives. Sometimes additional family members are also enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2000-11-07 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Identifying the change in the genetic information that causes recurrent hydatidiform moles. | Through study completion, an average of 15 years.
  The researchers will isolate genetic material from blood of women with recurrent hydatidiform molar (RHM) pregnancies, their RHM pregnancies, and for some first-degree relatives. DNA sequencing along with bioinformatic analysis will be used to find changes in the genetic code unique to individuals with RHM. When a new gene is found that shows variants that are deleterious to its function in at least 3 unrelated women with RHM, but not in healthy pregnant women, the outcome (finding a new genetic cause of RHM) will be achieved. RHM are very rare and only 70% have a known cause (known gene), thus the researchers will continue recruitment and enrollment of rare undiagnosed individuals when they are referred to the study. A key finding in one individual can provide the clue for a new disease gene in others. It cannot be predicted when this will happen, thus enrollment and data collection will continue as long as the protocol is open.
Identifying the changes in the genetic information that cause different forms of unexplained reproductive failure | Through study completion, an average of 15 years.
  The researchers will isolate genetic material from blood of women with recurrent unexplained reproductive failure (RF), their miscarried pregnancies if possible, and for some from first-degree relatives. DNA sequencing and bioinformatic analysis will be used to find changes in the genetic code unique to individuals with unexplained RF. When a new gene is found that shows variants that are deleterious to its function in at least 3 unrelated women with unexplained RF, but not in healthy pregnant women, the outcome (finding a new genetic cause for RF) will be achieved. Unexplained RF is relatively rare and many causes are not yet known, thus the researchers will continue recruitment and enrollment of rare undiagnosed individuals when they are referred to the study. A key finding in one individual can provide the clue for a new disease gene in others. It cannot be predicted when this will happen, thus enrollment and data collection will continue as long as the protocol is open

CONTACTS AND LOCATIONS:
Overall Officials: Ignatia B Van den Veyver, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The study is aimed to find the genetic cause of a rare condition, hydatidiform moles. Patient data with no identifying information will be published in aggregate following peer review in journals and/or presented at scientific meetings.
Supporting Information: Study Protocol
Time Frame: At the end of the study or when there is a new genetic finding
Access Criteria: Patient data with all identification removed will be published following peer review in journals and/or presented at scientific meetings.
  Reasonable requests from other researchers working on the same disease will be reviewed by the PI and sharing will be done after full deidentification and with institutionally approved of data and material transfer agreements.

REFERENCES:
- [Background] Kou YC, Shao L, Peng HH, Rosetta R, del Gaudio D, Wagner AF, Al-Hussaini TK, Van den Veyver IB. A recurrent intragenic genomic duplication, other novel mutations in NLRP7 and imprinting defects in recurrent biparental hydatidiform moles. Mol Hum Reprod. 2008 Jan;14(1):33-40. doi: 10.1093/molehr/gam079. Epub 2007 Nov 26. PMID 18039680
- [Background] Van den Veyver IB, Al-Hussaini TK. Biparental hydatidiform moles: a maternal effect mutation affecting imprinting in the offspring. Hum Reprod Update. 2006 May-Jun;12(3):233-42. doi: 10.1093/humupd/dmk005. Epub 2006 Mar 15. PMID 16540529
- [Background] Panichkul PC, Al-Hussaini TK, Sierra R, Kashork CD, Popek EJ, Stockton DW, Van den Veyver IB. Recurrent biparental hydatidiform mole: additional evidence for a 1.1-Mb locus in 19q13.4 and candidate gene analysis. J Soc Gynecol Investig. 2005 Jul;12(5):376-83. doi: 10.1016/j.jsgi.2005.02.011. PMID 15979551
- [Background] Al-Hussaini TK, Abd el-Aal DM, Van den Veyver IB. Recurrent pregnancy loss due to familial and non-familial habitual molar pregnancy. Int J Gynaecol Obstet. 2003 Nov;83(2):179-86. doi: 10.1016/s0020-7292(03)00209-1. PMID 14550593
- [Background] Saxena A, Frank D, Panichkul P, Van den Veyver IB, Tycko B, Thaker H. The product of the imprinted gene IPL marks human villous cytotrophoblast and is lost in complete hydatidiform mole. Placenta. 2003 Sep-Oct;24(8-9):835-42. doi: 10.1016/s0143-4004(03)00130-9. PMID 13129680
- [Background] Van den Veyver IB, Norman B, Tran CQ, Bourjac J, Slim R. The human homologue (PEG3) of the mouse paternally expressed gene 3 (Peg3) is maternally imprinted but not mutated in women with familial recurrent hydatidiform molar pregnancies. J Soc Gynecol Investig. 2001 Sep-Oct;8(5):305-13. doi: 10.1016/s1071-5576(01)00129-0. PMID 11677152
- [Background] Moglabey YB, Kircheisen R, Seoud M, El Mogharbel N, Van den Veyver I, Slim R. Genetic mapping of a maternal locus responsible for familial hydatidiform moles. Hum Mol Genet. 1999 Apr;8(4):667-71. doi: 10.1093/hmg/8.4.667. PMID 10072436
- [Background] Qian J, Deveault C, Bagga R, Xie X, Slim R. Women heterozygous for NALP7/NLRP7 mutations are at risk for reproductive wastage: report of two novel mutations. Hum Mutat. 2007 Jul;28(7):741. doi: 10.1002/humu.9498. PMID 17579354
- [Background] Slim R, Mehio A. The genetics of hydatidiform moles: new lights on an ancient disease. Clin Genet. 2007 Jan;71(1):25-34. doi: 10.1111/j.1399-0004.2006.00697.x. PMID 17204043
- [Background] Djuric U, El-Maarri O, Lamb B, Kuick R, Seoud M, Coullin P, Oldenburg J, Hanash S, Slim R. Familial molar tissues due to mutations in the inflammatory gene, NALP7, have normal postzygotic DNA methylation. Hum Genet. 2006 Oct;120(3):390-5. doi: 10.1007/s00439-006-0192-3. Epub 2006 Jul 28. PMID 16874523
- [Background] Murdoch S, Djuric U, Mazhar B, Seoud M, Khan R, Kuick R, Bagga R, Kircheisen R, Ao A, Ratti B, Hanash S, Rouleau GA, Slim R. Mutations in NALP7 cause recurrent hydatidiform moles and reproductive wastage in humans. Nat Genet. 2006 Mar;38(3):300-2. doi: 10.1038/ng1740. Epub 2006 Feb 5. PMID 16462743
- [Background] Fisher RA, Hodges MD, Newlands ES. Familial recurrent hydatidiform mole: a review. J Reprod Med. 2004 Aug;49(8):595-601. PMID 15457849
- [Background] Zhao J, Moss J, Sebire NJ, Cui QC, Seckl MJ, Xiang Y, Fisher RA. Analysis of the chromosomal region 19q13.4 in two Chinese families with recurrent hydatidiform mole. Hum Reprod. 2006 Feb;21(2):536-41. doi: 10.1093/humrep/dei357. Epub 2005 Oct 20. PMID 16239310
- [Background] Fisher RA, Hodges MD, Rees HC, Sebire NJ, Seckl MJ, Newlands ES, Genest DR, Castrillon DH. The maternally transcribed gene p57(KIP2) (CDNK1C) is abnormally expressed in both androgenetic and biparental complete hydatidiform moles. Hum Mol Genet. 2002 Dec 15;11(26):3267-72. doi: 10.1093/hmg/11.26.3267. PMID 12471053
- [Background] van der Smagt JJ, Scheenjes E, Kremer JA, Hennekam FA, Fisher RA. Heterogeneity in the origin of recurrent complete hydatidiform moles: not all women with multiple molar pregnancies have biparental moles. BJOG. 2006 Jun;113(6):725-8. doi: 10.1111/j.1471-0528.2006.00929.x. PMID 16709217
- [Background] Mahadevan S, Wen S, Balasa A, Fruhman G, Mateus J, Wagner A, Al-Hussaini T, Van den Veyver IB. No evidence for mutations in NLRP7 and KHDC3L in women with androgenetic hydatidiform moles. Prenat Diagn. 2013 Dec;33(13):1242-7. doi: 10.1002/pd.4239. Epub 2013 Oct 4. PMID 24105752
- [Background] Mahadevan S, Wen S, Wan YW, Peng HH, Otta S, Liu Z, Iacovino M, Mahen EM, Kyba M, Sadikovic B, Van den Veyver IB. NLRP7 affects trophoblast lineage differentiation, binds to overexpressed YY1 and alters CpG methylation. Hum Mol Genet. 2014 Feb 1;23(3):706-16. doi: 10.1093/hmg/ddt457. Epub 2013 Sep 18. PMID 24105472